CLINICAL TRIAL: NCT06925074
Title: Quantified Evaluation of Noninvasive System Delivering Microwave Energy for Unwanted Fat Reduction and Skin Tightening in Asians.
Status: Not yet recruiting | Type: Observational
Sponsor: Chang Chang Cheng (Other)
Collaborators: GRAND Medical Co., Ltd. (Unknown)
Responsible Party: Sponsor-Investigator, Chang Chang Cheng, Associate Professor, China Medical University Hospital
Organization: China Medical University Hospital (Other)
Other Study IDs: CMUH114-REC2-040
Record Dates: First submitted 2025-04-06; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Facial Aging; Skin Laxity; Cheek Wrinkles
Keywords: 3D imaging; Skin laxity; Microwaves; Fat reduction; Facial aging
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to evaluate the effectiveness and safety of microwave-assisted heating technology in facial fat reduction and skin tightening in Asians.

The main questions it aims to answer are:

1. How effective is the microwave-based system in reducing fat and tightening Skin?
2. What objective methods can be used to measure treatment outcomes?
3. What are the optimal treatment parameters for maximum efficacy?
4. What are the safety and side effects associated with the treatment?
5. How long-lasting are the results?

Participants will go through three treatment sessions using the "DEKA" ONDA Microwave treatment system, with each session lasting 12 minutes.

DETAILED DESCRIPTION:
As people age, facial skin sagging and submental fat accumulation have become concerns for many, not only affecting their appearance but also negatively impacting their self-confidence. With the continuous advancement of modern medical aesthetic technology, noninvasive treatments like microwave-assisted heating technology have provided new solutions for addressing these issues.

The microwave-assisted heating technology works by precisely heating subcutaneous fat tissue with high-frequency energy, inducing fat cell apoptosis while simultaneously stimulating collagen production in the skin, thereby achieving fat reduction and skin tightening. Compared to traditional surgical methods, this technique offers the advantages of being non-invasive, having a short recovery period, and carrying lower risks.

To further investigate these effects, we plan to conduct a prospective, open-label clinical trial. The treatment will focus on enhancing the mid and lower facial area, while carefully managing the treatment time and monitoring patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 20 and 60.
* Subjects who are capable of understanding and comply with the study procedures, instructions, and visit schedule.
* Subjects who voluntarily decide to participate in the entire course of the trial and provide written consent in the Informed Consent Form.

Exclusion Criteria:

* Subjects with autoimmune diseases/received immunotherapy and subjects with diabetes mellitus.
* Subjects with a history of a hypertrophic scar.
* Pregnant or breastfeeding women.
* Subjects with untreated epilepsy or underlying porphyria.
* When there is an active disease (such as inflammation, infection or tumors) in or near the intended treatment site.
* Treatment procedure (e.g., bioresorbable fillers, laser/light therapies, botulinum toxin A injections, facial lift, facial peels, excisional facial surgery, dermal photorejuvenation, oral or maxillofacial surgery, etc.) that may interfere with the treatment area or evaluation within 6 months before screening as determined by the Principal Investigator.
* The subject who received soft tissue augmentation at the treatment site at any time before screening as determined by the Principal Investigator.
* Subjects with a scar or skin lesion at the treatment site that may interfere with the judgment of the treatment effect.
* Subjects who participated in another clinical trial within 60 days before screening or plan to participate in another investigation during this study.
* Subjects who plan to receive other wrinkle improvement treatments in the face during this trial.
* Subjects who are otherwise determined by the investigator as ineligible for this study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Men and women aged between 20 and 60.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Eyebrow Peak angle | At week 0, 4, 12
  The vertices of the Eyebrow Peak angles lie at the static point eyebrow head, measured against a horizontal line parallel to the ground.
Eyebrow Tail angle | At week 0, 4, 12
  The vertices of the Eyebrow Tail angles lie at the static point eyebrow head, measured against a horizontal line parallel to the ground.
Pupil-Eyebrow Peak angle | At week 0, 4, 12
  The Pupil-Eyebrow Peak angle is then measured between this line and another line connecting nasal to eyebrow peak.
Canthus-Oral-Nasal angle | At week 0, 4, 12
  The Canthus-Oral-Nasal angle is measured between a line connecting oral commissure to nasal and a line connecting oral commissure to lateral canthus.
Eyebrow-Orbital length | At week 0, 4, 12
  The linear distances from point superior orbital rim to the inferior border of eyebrow.
Orbital-Upper Eyelid length | At week 0, 4, 12
  The linear distances from point superior orbital rim to the superior border of palpebral fissure.
Vertical Palpebral Fissure length | At week 0, 4, 12
  The size of the palpebral fissure can be determined by measuring the vertical distance between the superior and inferior borders of palpebral fissure when the eyes are at rest.
Eyebrow-Iris length | At week 0, 4, 12
  The horizontal distance between the lateral limbus of the iris and the eyebrow peak .
Tragus-Oral length | At week 0, 4, 12
  The distances between the bilateral tragi passing through the oral commissure.
Lower Facial Contouring length | At week 0, 4, 12
  The distances between the bilateral tragi passing through the mental protuberance.
Antiaging Scales for facial rejuvenation | At week 0, 4, 12
  A table that shows the antiaging scale system utilizing the 4 angular and 6 linear measurements described above. Index 5 is identified as "neutral" or "no significant changes". Total score for the whole face was 100; either lower or higher than 50 suggesting "aging" or "rejuvenation, respectively".
  °: degree; mm: millimeter.
LifeViz® Mini 3D imaging system | At week 0, 4, 12
  This 3D photographic system can be used to calculate the differences in volume in a treated area precisely and accurately for professional patient follow-up.

SECONDARY OUTCOMES:
Global Aesthetic lmprovement Scale | At week 0, 2, 4, 12
  -1: Worse. Appearance worse than the original condition or with complications. 0: No change. Appearance essentially the same as the original condition.
  1. Improved. Obvious improvement, but touch-up or re-treatment is indicated.
  2. Much Improved. Marked improvement in the condition, but not optimal for the patient; a touch-up would slightly improve the outcome
  3. Very much improved. Optimal cosmetic result for the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taichung, Taiwan

REFERENCES:
- [Background] Salsi B, Fusco I. Non-invasive system delivering microwaves energy for unwanted fat reduction and submental skin tightening: Clinical evidence. J Cosmet Dermatol. 2022 Nov;21(11):5657-5664. doi: 10.1111/jocd.15205. Epub 2022 Jul 19. PMID 35778895
- [Background] Spiroski M. Retraction: Five papers from Open Access Maced J Med Sci. Vol. 7 No. 18 (2019): Sep 30 (Global Dermatology). Open Access Maced J Med Sci. 2020 Sep 30;8(B):573. doi: 10.3889/oamjms.2020.5492. PMID 32996903